CLINICAL TRIAL: NCT04653077
Title: Bone Marrow Stem Cells Transplantation for the Treatment of Cerebral Palsy
Brief Title: MSCs Therapy for Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aljazeera Hospital (Other)
Collaborators: AMR KHALIL ORTHOPEDIC SURGERY CENTER (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: cerebral palsy
Record Dates: First submitted 2020-11-27; First posted 2020-12-04 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-11

CONDITIONS: Stem Cell Transplant Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- stem cells (Experimental): Intravenous and Intrathecal transplantation of specific populations of purified bone marrow-derived stem cells and mesenchymal stem cells.
  Interventions: Other: stem cells

INTERVENTIONS:
Other: stem cells — Intravenous and Intrathecal transplantation of specific populations of purified bone marrow-derived stem cells and mesenchymal stem cells.

SUMMARY:
Cerebral palsy (CP) is the most common physical disability in childhood. CP comprises a heterogeneous group of disorders that are the result of a non-progressive disruption or injury that occurred during fetal brain development or within the first two years of life.

DETAILED DESCRIPTION:
This disruption can result in spasticity, dystonia, muscle contractures, weakness and difficulty in coordination that ultimately affects the ability to control movements. Resultant activity limitations may affect gross motor movements, fine motor movements, speech and communication, as well as eating and drinking.

ELIGIBILITY:
Inclusion Criteria:

* • Must be more than 2 year of age and less than 12 years of age at the time of screening for inclusion in the study.

  * Clinical evidence of a non-progressive motor disability due to brain dysfunction.

Exclusion Criteria:

* • Intractable seizures

  * Traumatic brain injury
  * Genetic disorder
  * Current Infection
  * Renal insufficiency
  * Hepatic disease
  * HIV+ (as demonstrated by positive blood test)
  * Immunosuppression

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2020-12-02 (Estimated); Primary Completion 2022-10-15 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Motor Performance. | 6 months
  the number of patients who will have changes in motor performance

CONTACTS AND LOCATIONS:
Locations (1):
- Aljazeera( Al Gazeera) hospital, Giza, Egypt